CLINICAL TRIAL: NCT03079895
Title: The Thrive Care Study: Computer-Delivered Cognitive Behavioral Therapy as Care Augmentation for Depressed Primary Care Patients
Brief Title: Thrive Care: Internet CBT for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KP-RRC-20150408
Record Dates: First submitted 2017-02-01; First posted 2017-03-15 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Depression; internet; Cognitive Behavioral Therapy; CBT; computer; Primary Care; Psychiatry; treatment; self-help; managed care
MeSH Terms: conditions — Depression | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Control arm will receive treatment as usual for depression from primary care physician. Intervention arm will also receive treatment as usual, and access to an internet-based self-help tool for treatment of depression, along with coaching emails and/or phone calls, encouraging their participation and answering questions about how to use the program.
Who Masked: Care Provider
Masking Description: The primary care physician will not receive feedback about which arm the patient was assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): After enrollment in the study, the subject will continue to receive treatment as usual for their depression from their primary care physician. They then will be asked to complete 2-month and 6-month assessments about their emotional well-being.
- Intervention Arm (Experimental): After enrollment in the study, the subject will be granted 8 weeks of access to "Thrive", an online self-help tool designed to assess for depressive symptoms and give therapeutic suggestions based on Cognitive Behavioral Therapy. During the first 4 weeks, they will receive 4 coaching emails and/or phone calls encouraging their participation in the study, and answering any program-related questions. The subject will also continue to receive treatment as usual for their depression from their primary care physician. They then will be asked to complete 2-month and 6-month assessments about their emotional well-being.
  Interventions: Behavioral: Thrive

INTERVENTIONS:
Behavioral: Thrive — Thrive is an online self-help tool designed to assess for depressive symptoms and give therapeutic suggestions based on Cognitive Behavioral Therapy principals.
  Other Names: Thrive for Depression
  Arms: Intervention Arm

SUMMARY:
This project will study the effectiveness of computerized cognitive behavioral therapy (CBT) in reducing depression symptoms. The design is a two-arm randomized controlled trial comparing (i) control arm, which is treatment as usual with (ii) treatment arm, which is treatment as usual plus computerized CBT. The primary outcome measure is change in depression symptom severity. The name of the computerized CBT program to be used in the study is Thrive.

DETAILED DESCRIPTION:
Population:

* As identified in Epic, Kaiser Permanente Southern California (KPSC) Fontana Family Medicine patients with a depression diagnosis recorded during the prior week (rolling basis).
* Target study enrollment: 150 participants per arm (300 total)

Recruitment:

* Kaiser Permanente (KP) will send eligible patients a postal letter inviting them to participate in study. Interested patients will be directed to the Enrollment/Assessment Website, a website to be developed by vendor Waypoint Health Innovations. The recruitment letter will contain (i) a description of the study, (ii) the web address for the Enrollment/Assessment Website, (iii) the patient's Study Identifier (ID).
* Additionally, KP will send eligible patients for whom KP has an email address an email inviting them to participate in the study.

Screening and Enrollment (Enrollment/Assessment Website):

* A patient interested in applying to the study will visit the Enrollment/Assessment Website and input his/her unique Study ID. The website will verify that the entered Study ID is on a pre-loaded list. If valid, the patient may continue to screening assessments.
* Patient will complete the 9-item Patient Health Questionnaire (PHQ-9) depression symptom assessment. Patients with eligible PHQ-9 scores may continue to Informed Consent page.
* The Informed Consent (IC) page will contain (i) the Informed Consent text including contact information for any questions patient may have; (ii) fields for first name, last name, date of birth, email address, and phone number; (iii) a check box labeled "I understand the above information and agree to participate…" (or similar); and (iv) a "submit" (or similar) button.
* To enroll in the study, the patient must complete all fields, check the box, and click submit button. The website will validate that every field has been completed and that the phone number and email fields have the correct format (e.g. name@domain.com for the email field).
* If all fields are complete, the website will store the Study ID, first name, last name, date of birth, email address, and phone number that patient entered into the website. They will be stored in an encrypted database for use by researchers.
* Additionally, the website will store the complete Informed Consent page (including Informed Consent text, first name, last name, date of birth, email address, phone number, and checked box) in a single encrypted record, timestamp it, and place a digital certificate on it. The digital certificate will allow us to prove that no one tampered with any part of the IC document after the participant clicked submit.
* The website automatically randomizes participants to treatment or control arm. Participants continue in website to baseline assessments.
* After baseline assessments, control arm participants go to a page in the Enrollment/Assessment Website telling them to expect assessment again in 2 months, while treatment arm participants will be given instructions for enrolling in Thrive.
* Researchers would have access to the completed IC forms to print and/or mail to patients who request a copy.
* Weekly, KP research coordinator will review new participants' study ID, name, and date of birth (DOB) the participant entered to ensure they match KP records. Individuals who entered information that does not reasonably match KP records would be removed from the study.

Coaching:

• KP will send each treatment arm participant four emails encouraging them to use Thrive, with the exception that the second email will be replaced by a phone call from KP for patients who have not achieved a minimum level of activity in Thrive at that point.

Endpoint and Follow-up Assessments:

• KP will ask each study participant to visit Enrollment/Assessment Website 2 and 6 months after study enrollment to complete assessments.

ELIGIBILITY:
Inclusion Criteria:

* Per EPIC (or other system) records, clinical depression was addressed during the prior week by a KPSC Fontana Family Medicine physician , reflected by an ICD-9 or ICD-10 diagnosis of Depression, Major Depressive Disorder, Dysthymia, Adjustment Disorder with Depressed Mood, and Depression Not Otherwise Specified. This does not have to be the patient's first depression diagnosis.
* Screening Patient Health Questionnaire (PHQ-9) score of ≥5 as measured in Assessment Website (see Section 4 for information on Assessment Website)

Exclusion Criteria:

* History or current diagnosis indicating any Schizophrenia spectrum or other psychotic disorder, any Neurocognitive disorder, Delirium, Bipolar disorder, Intellectual disability, or Personality disorder, or any active substance abuse, as defined by DSM-5
* Member is not proficient in English
* Member answered "more than half the days" or "nearly every day" on the Patient Health Questionnaire ninth item and did not subsequently answer (regarding suicidal ideations) "Yes" to the question "are you sure you can stay safe?"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
PHQ-9 score change | 0-6 months after enrollment
  Change in score on the 9-item Patient Health Questionnaire

SECONDARY OUTCOMES:
GAD-7 score change | 0-6 months after enrollment
  Change in score on 7-item Generalized Anxiety Disorder scale
Quality of Life change | 0-6 months after enrollment
  Change in subjective measure of subject's quality of life (based on Behavioral Risk Factor Surveillance System)
Workplace productivity change | 0-6 months after enrollment
  Change in subjective measure of subject's workplace productivity (based on Behavioral Risk Factor Surveillance System)
Medication adherence | 0-6 months after enrollment
  Measure of compliance with prescribed medications, based on a single item question
Psychotherapy utilization | 12 months prior to enrollment, through 6 months after enrollment
  Subjective measurement of whether or not the subject has received psychotherapy from a licensed provider
Psychiatric specialty utilization | 0-6 months after enrollment
  Subjective measurement of whether or not the subject has received treatment from a provider in the Department of Psychiatry
Satisfaction with Thrive | 2 months after enrollment
  Subjective measurement of how satisfied patient was with the treatment intervention
Satisfaction with Kaiser Permanente Southern California | 0-6 months after enrollment
  Subjective measurement of how satisfied patient was with their experience of care at Kaiser Permanente Southern California
Thrive Adherence | 0-2 months after enrollment
  Percent enrolled in Thrive over total number invited, number of logins and lessons started

CONTACTS AND LOCATIONS:
Overall Officials: Roderick R Stuart, MD, Principal Investigator — Southern California Permanente Medical Group
Locations (1):
- Kaiser Fontana Medical Center, Fontana, California, United States

IPD SHARING:
Plan to Share IPD: No